CLINICAL TRIAL: NCT05384600
Title: Incisional Hernia Prevention: Risk-benefit From a Patient's Perspective
Acronym: INVITE
Status: Completed | Type: Observational
Sponsor: Cardiff and Vale University Health Board (Other Government)
Responsible Party: Sponsor
Other Study IDs: 8342; 310695 (Registry Identifier: IRAS)
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2022-07

CONDITIONS: Incisional Hernia
Keywords: Surgical Mesh; Acceptability; Prevention; Qualitative Research
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with Incisional Hernia: Patients who have undergone elective or emergency colonic resection between 2017 and 2020 at Cardiff and Vale UHB, who have subsequently received a diagnosis of Incisional Hernia. One-off self-completed patient questionnaire upon enrolment. Sub-set will be invited to participant in qualitative interview.
- Patients without Incisional Hernia: Patients who have undergone elective or emergency colonic resection between 2017 and 2020 at Cardiff and Vale UHB, who have not subsequently been diagnosed with (or suspected of having) incisional hernia. One-off self-completed patient questionnaire upon enrolment. Sub-set will be invited to participant in qualitative interview.
- Patients due to undergo surgery: Patients who are due to undergo elective colonic surgery within Cardiff and Vale UHB, who have an unknown risk of- , and may or may not go on to develop-, incisional hernia. One-off self-completed patient questionnaire upon enrolment. Sub-set will be invited to participant in qualitative interview.

SUMMARY:
Incisional Hernia (IH) is a common complication of abdominal surgery and causes serious morbidity to patients. IH formation is multifactorial and its risk varies from patient to patient. Risk-predictive tools have been developed to identify patients at high risk of IH before their initial operation, with high-risk patients possibly being offered the use of prophylactic mesh, placed at the end of the operation to prevent IH from forming. With controversy surrounding the use of mesh in other types of surgery, however, it is not known if mesh use is acceptable to patients. This study aims to assess how patients feel about prophylactic mesh and whether it is acceptable to them.

DETAILED DESCRIPTION:
Incisional hernias are bulges through the abdominal wall that occur at the site of previous surgery. They are common, affecting between 12-20% of patients undergoing abdominal surgery, can pose a significant cost to the NHS and cause serious morbidity to patients.

Risk-prediction tools are being developed with the aim of working out a person's risk of developing an incisional hernia before their operation. It is hoped that this will allow surgeons to give patients an idea of what their risk is before the operation happens so that patients can understand if they are at high, medium or low risk, and what they might be able to do about it before the operation.

For patients that are "high risk" for developing an incisional hernia, it may be possible to use a synthetic mesh, similar to those used to fix groin hernias. This would be placed in the wound at the end of the initial operation to strengthen the wound to try and reduce the chance of developing an incisional hernia, however to date, no studies have looked at whether patients would find this acceptable.

This study aims to establish whether mesh placed to prevent hernias during the initial surgery would be acceptable to patients. This, in turn, can be used to inform the design of future research studies surrounding the use of surgical mesh.

ELIGIBILITY:
Inclusion Criteria:

Group 1 Patients who have previously undergone abdominal surgery, and subsequently developed incisional hernia.

* Over the age of 18 years old
* Able and willing to provide valid informed consent
* Undergone elective or emergency colonic resection >12 months ago
* Clinical or radiological diagnosis of incisional hernia.

Where possible, patients will only be approached to participate where their clinical record indicates they are aware that they have a diagnosis of incisional hernia.

Group 2 Patients who have undergone abdominal surgery, but have not subsequently developed incisional hernia.

* Over the age of 18 years old
* Able and willing to provide valid informed consent
* Undergone emergency abdominal surgery > 12 months ago OR elective colonic resection > 12 months ago
* Do not have a clinical or radiological diagnosis of Incisional hernia (or suspected incisional hernia)

Group 3 Patients who are due to undergo abdominal surgery, who may or may not subsequently develop incisional hernia.

* Over the age of 18 years old
* Able and willing to provide valid informed consent
* Scheduled for elective colonic resection in Cardiff and Vale UHB.
* No history of previous laparotomy.

Where possible, attempts will be made to identify patients undergoing colonic resection for benign disease.

Exclusion Criteria:

All participants (groups 1, 2 & 3)

* Unable or unwilling to give informed consent
* Palliative diagnosis either at time of surgery, or since
* Inability to understand or complete study questionnaires, due to intellectual or cognitive impairment or due to insufficient English-language skills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In order to explore patient perceptions of surgical mesh use in the context of incisional hernia prevention, we will identify three groups of patients, from the department of surgery, Cardiff and Vale University Health Board:
  1. Patients that have previously undergone abdominal surgery and subsequently been diagnosed with incisional hernia. (n=150)
  2. Patients that have previously undergone abdominal surgery and have not subsequently developed or been diagnosed with incisional hernia. (n=150)
  3. Patients that are currently due to undergo abdominal surgery, and may or may not subsequently develop incisional hernia. (n=20)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Acceptability of prophylactic surgical mesh use to patients | 12 months
  A combination of qualitative and quantitative methods will explore patient perceptions of prophylactic mesh. Non-validated questionnaire developed based on Health Belief Model Theory, consisting of multiple 5-point Likert scale (min.1, max. 5), used in combination with semi-structured interviews to evaluate:
  A) Understanding of surgical mesh B) Perceptions of surgical mesh risk C) Perceptions of surgical mesh benefit
Impact of incisional hernia risk scores on surgical mesh acceptibility | 12 months
  A combination of qualitative and quantitative methods will explore how incisional hernia risk impacts perception of surgical mesh use
  Non-validated questionnaire developed based on Health Belief Model Theory, consisting of multiple 5-point Likert scale (min.1, max. 5), used in combination with semi-structured interviews to evaluate:
  A) Perception of risk in relation to incisional hernia B) Perception of personalised risk scoring C) Impact of A) and B) on surgical mesh use

SECONDARY OUTCOMES:
Patient understanding of Incisional Hernia | 9 months
  Patient-reported understanding of incisional hernia will be assessed using non-validated questionnaire, developed based on the Health Belief Model Theory. Multiple 5-point Likert scale questions, where 1 (min.) represents least perceived understanding possible and 5 (max.) represents most perceived understanding possible.
Factors that modify acceptability of surgical mesh | 9 months
  Semi-structured interviews will use qualitative research techniques to explore factors that impact patient acceptability of surgical mesh .

CONTACTS AND LOCATIONS:
Overall Officials: Julie Cornish, Principal Investigator — Cardiff and Vale University Health Board
Locations (1):
- Julie Cornish, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith L, Meggy A, Watts T, Knight L, Torkington J, Cornish J. Incisional hernia prevention: risk-benefit from a patient perspective (INVITE) - protocol for a single-centre, mixed-methods, cross-sectional study aiming to determine if using prophylactic mesh in incisional hernia prevention is acceptable to patients. BMJ Open. 2022 Dec 30;12(12):e069568. doi: 10.1136/bmjopen-2022-069568. PMID 36585153